CLINICAL TRIAL: NCT01684319
Title: Prospective, Randomized, Double Blind and Placebo Controlled Study With the Aim to Establish the Role of Milk Proteins in Gastrointestinal Diseases (GERD, Constipation and Colics) of Young Infants and to Determine the Diagnostic Value of Immunological Tests in These Pathologies.
Brief Title: Milk-induced Gastrointestinal Symptoms in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Philippe Eigenmann, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 11-202 (MATPED 11-047)
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Gastrointestinal Symptoms in Young Infants
Keywords: Constipation; Gastroeosphageal reflux; Colics
MeSH Terms: conditions — Constipation; Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infant formula milk (Placebo Comparator): Infant formula milk adapted to age of infant
  Interventions: Dietary Supplement: Placebo
- Formula milk free of milk proteins (Active Comparator): Milk-free formula milk adapted to age of infant
  Interventions: Dietary Supplement: Formula milk free of cow's milk protein

INTERVENTIONS:
Dietary Supplement: Formula milk free of cow's milk protein
  Arms: Formula milk free of milk proteins
Dietary Supplement: Placebo — Infant formula milk
  Arms: Infant formula milk

SUMMARY:
Various digestive manifestations are common in infants less than 6 months and have a significant impact on morbidity and quality of life of the family. In a prospective study on more than 2800 Italian infants followed by 0-6 months of life, it was determined that 55% of these children had gastrointestinal symptoms such as regurgitation (23%), colics (20%), constipation (17%) or poor weight gain (15%). However, these symptoms are not very accurate, and their cause is often difficult to determine. Frequently, the pediatrician will exclude cow's milk protein in infant feeding, but without a clear etiological diagnosis was asked. This measure causes significant additional costs through the use of extensively hydrolyzed milk specifically for children and involves an elimination diet of all foods containing cow's milk sometimes for several years. This can negatively influence the growth of the child.

If the involvement of milk in these pathologies is suggested by some early studies (35% for colics, 68% in constipation, 42% in gastroesophageal reflux), it is unclear in the current state of knowledge if these gastrointestinal symptoms are actually due to an "allergy" to milk. Moreover, there is no validated diagnostic test for non-IgE-mediated gut allergy. However, various tests have proven their effectiveness in the investigation of non IgE-mediated allergy (eg. LAT, patch tests) and will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Infants 0-6 month old with at least one of the following symptoms : constipation, gastroesophageal reflux, colics

Exclusion Criteria:

* Prematurity
* exclusive breastfeeding
* Other cause for symptoms

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Milk allergy in gastrointestinal diseases in young infants | 10 weeks
  Establish the role of milk proteins in gastrointestinal diseases in young infants

SECONDARY OUTCOMES:
Diagnostic tests | 10 weeks
  Determine the diagnostic value of immunological tests in these pathologies

CONTACTS AND LOCATIONS:
Overall Officials: Philippe A Eigenmann, MD, Study Director — Hôpitaux Unversitaire de Genève
Locations (1):
- Département de l'enfant et de l'adolesent - Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland